CLINICAL TRIAL: NCT04852484
Title: Morphine Versus Ketamine as Adjuvants in Ultrasound-guided Paravertebral Thoracic Blocks in Elective Thoracic Surgery
Brief Title: Morphine Versus Ketamine as Adjuvants in Paravertebral Blocks
Acronym: Annie-Dimitr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aretaieion University Hospital (Other)
Collaborators: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 307/26-03-2021
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Pain, Neuropathic; Morphine; Ketamine; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Neuralgia; Agnosia | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- local anesthetic and morphine group (Active Comparator): paravertebral block with local anesthetic and morphine, followed by a continuous infusion of local anesthetic and morphine in the paravertebral space
  Interventions: Drug: local anesthetic-morphine
- local anesthetic and ketamine group (Active Comparator): paravertebral block with local anesthetic and ketamine, followed by a continuous infusion of local anesthetic and ketamine in the paravertebral space
  Interventions: Drug: local anesthetic-ketamine
- local anesthetic group (Active Comparator): paravertebral block with local anesthetic only, followed by a continuous infusion of local anesthetic only in the paravertebral space
  Interventions: Drug: local anesthetic

INTERVENTIONS:
Drug: local anesthetic-morphine — Before the operation, 19 mL of 0.5% Ropivacaine + 2 mg of morphine (20 mL in total) will be injected in the paravertebral space. Afterwards, there will be a pump of 500 ml of 0.2 % ropivacaine + 6 mg of morphine connected to the catheter after the end of the surgery, administered continuously at a rate of 10 mL/hr
  Other Names: local anesthetic and morphine administered paravertebrally
  Arms: local anesthetic and morphine group
Drug: local anesthetic-ketamine — Before the operation, 19 mL of 0.5% Ropivacaine + 50 mg of ketamine (20 mL in total) will be injected in the paravertebral space. Afterwards, there will be a pump of 500 ml of 0.2 % ropivacaine + 200 mg of ketamine connected to the catheter after the end of the surgery, administered continuously at a rate of 10 mL/hr
  Other Names: local anesthetic and ketamine administered paravertebrally
  Arms: local anesthetic and ketamine group
Drug: local anesthetic — Before the operation, 19 mL of 0.5% Ropivacaine + 1 mL of normal saline (20 mL in total) will be injected in the paravertebral space. Afterwards, there will be a pump of 500 ml of 0.2 % ropivacaine connected to the catheter after the end of the surgery, administered continuously at a rate of 10 mL/hr
  Other Names: local anesthetic administered paravertebrally
  Arms: local anesthetic group

SUMMARY:
The aim of this study will be to compare the effects of morphine versus ketamine when they are used as adjuvants to the local anesthetic in paravertebral nerve blocks performed with the aid of ultrasound. Furthermore, a group of local anesthetic without an adjuvant, will also be compared to the two groups

DETAILED DESCRIPTION:
Elective thoracotomies are usually performed for removal of pathological masses in the mediastinum, lung parenchyma and upper gastrointestinal system. They are considered to be painful operations, related to both acute and chronic pain (post- thoracotomy pain syndrome), the latter lasting for a minimum period of 2 months.

Post-operative thoracic pain is associated often with diaphragmatic dysfunction, which can also lead to atelectasis and pneumonia and post-operative pulmonary complications in general.

Several techniques have been tried in order to minimize such events. Thoracic epidural analgesia, intravenous analgesia, intercostal blocks, local infiltration of local anesthetics by the surgeon are some of them.

Paravertebral thoracic blocks have become increasingly popular in recent years since they are less likely to cause neurologic complications than thoracic epidural analgesia. Moreover, bleeding disorders, and use of anti-coagulant and anti- thrombotic medications, which are considered as contraindications to an epidural procedure, are not strict contraindications in the performance of paravertebral blocks, especially when they are performed under ultrasonographic guidance.

Ropivacaine and Levobupivacaine are the most popular local anesthetics that have been used. Moreover, several adjuvants have been added to them in order to enhance the effects of those blocks. Dexamethasone, Morphine, Dexmedetomidine, Clonidine, Ketamine, Magnesium Sulphate are some of them. Results are variable.

The rationale behind adjuvants used to enhance effects of local anesthetics is the fact that some seem to act directly in the spinal cord receptors and the central nervous system. The effect of morphine on the dorsal horns of the spinal cord has been extensively studied in the past. Due to its limited lipophilicity, it is assumed that administering the specific drug to the paravertebral space could lead to its transfer and action on the dorsal horns.

On the other hand, the action of ketamine seems to be by blocking N-Methyl-D-Aspartate (NMDA) receptors in the spinal cord. It is also considered to have an effect on voltage sensitive Ca2+ channels, opioid receptors, and monoaminergic receptors. Therefore, it is considered overall to affect nociception.

Overall, it is assumed that morphine might have an effect on the dorsal horns of the spinal cord, and ketamine on NMDA receptors at "higher pain centers". It is also assumed that there will be some degree of systemic absorption due to the rich vascular supply of the specific area. The investigators aim to compare the effects of those two when they are used as adjuvants to the local anesthetic in paravertebral nerve blocks performed with the aid of ultrasound. Furthermore, a group of local anesthetic without an adjuvant, will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective thoracotomy for any cause
* American Society of Anesthesiologists class I-III (ASA I-III)

Exclusion Criteria:

* known allergy to local anesthetic
* local inflammation
* paravertebral tumor
* severe respiratory distress ( breathing dependence on accessory muscles)
* severe spinal deformities
* severe ipsilateral diaphragmatic paresis
* morbid obesity (BMI>35 kg/m2)
* blood coagulation disorders
* known contraindication for administration of ketamine or morphine
* psychiatric disorders
* severe cardiovascular disease
* systematic use of opioids due to chronic pain
* renal or hepatic failure
* patients who refuse to participate

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
morphine consumption in the first 48 hours | 48 hours postoperatively
  patients will be followed for cumulative morphine consumption through patient-controlled analgesia device for 48 hours postoperatively

SECONDARY OUTCOMES:
morphine consumption in Post-Anesthesia Care Unit (PACU) | 24 hours postoperatively
  mg of morphine requested during patient PACU stay
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 12 hours postoperatively | 12 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 12 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 48 hours postoperatively | 48 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 48 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
morphine consumption in the first 6 hours | 6 hours postoperatively
  patients will be followed for cumulative morphine consumption through patient-controlled analgesia device for 6 hours postoperatively
morphine consumption in the first 12 hours | 12 hours postoperatively
  patients will be followed for cumulative morphine consumption through patient-controlled analgesia device for 12 hours postoperatively
morphine consumption in the first 24 hours | 24 hours postoperatively
  patients will be followed for cumulative morphine consumption through patient-controlled analgesia device for 24 hours postoperatively
side effects postoperatively | 96 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively
satisfaction from postoperative analgesia | 48 hours postoperatively
  satisfaction from postoperative analgesia on a four-point Likert scale with 1 marked as minimal satisfaction and 4 as maximal satisfaction
morphine requirement during surgery | intraoperatively
  dose of required morphine administered intraoperatively
time to first request for analgesia | during stay in Post-Anesthesia Care Unit, 24 hours postoperatively
  the time for the first patient request for analgesia will be noted
hospitalization time | 7 days postoperatively
  duration of hospital stay after surgery in days
incidence of chronic pain 3 months after surgery | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
incidence of chronic pain 6 months after surgery | 6 months after surgery
  occurrence of chronic pain at the site of the operation 6 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (2):
- Greece (2):
  - Aretaieion University Hospital, Athens
  - KAT General Hospital of Athens, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] El Mourad MB, Amer AF. Effects of adding dexamethasone or ketamine to bupivacaine for ultrasound-guided thoracic paravertebral block in patients undergoing modified radical mastectomy: A prospective randomized controlled study. Indian J Anaesth. 2018 Apr;62(4):285-291. doi: 10.4103/ija.IJA_791_17. PMID 29720754
- [Background] Ahmed MJ, Ur Rehman A, Arshad RM, Amjad MWA, Khan Z, Furqan A. Efficacy of Dexmedetomidine vs Morphine as an Adjunct in a Paravertebral Block with Bupivacaine in Postoperative Analgesia Following Modified Radical Mastectomy. Cureus. 2020 May 22;12(5):e8231. doi: 10.7759/cureus.8231. PMID 32582491
- [Background] Mao Y, Zuo Y, Mei B, Chen L, Liu X, Zhang Z, Gu E. Efficacy of perineural dexamethasone with ropivacaine in thoracic paravertebral block for postoperative analgesia in elective thoracotomy: a randomized, double-blind, placebo-controlled trial. J Pain Res. 2018 Sep 11;11:1811-1819. doi: 10.2147/JPR.S164225. eCollection 2018. PMID 30254483
- [Background] Maruyama Y, Shimoji K, Shimizu H, Sato Y, Kuribayashi H, Kaieda R. Effects of morphine of human spinal cord and peripheral nervous activities. Pain. 1980 Feb;8(1):63-73. doi: 10.1016/0304-3959(80)90090-1. PMID 7367037
- [Background] Kathirvel S, Sadhasivam S, Saxena A, Kannan TR, Ganjoo P. Effects of intrathecal ketamine added to bupivacaine for spinal anaesthesia. Anaesthesia. 2000 Sep;55(9):899-904. doi: 10.1046/j.1365-2044.2000.01472.x. PMID 10947756